CLINICAL TRIAL: NCT01945333
Title: Personalized and Scalable Cognitive Remediation Approaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Alice Medalia, Clinical Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #6721; 1R34MH100317-01 (NIH)
Record Dates: First submitted 2013-09-13; First posted 2013-09-18 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Cognitive remediation; Schizophrenia; Schizoaffective disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Brain Basics for Impaired Tone Matchers (Active Comparator): Cognitive remediation includes sensory processing training
  Interventions: Behavioral: Cognitive remediation
- Brain Basics for Intact Tone Matchers (Active Comparator): Cognitive remediation includes sensory processing training
  Interventions: Behavioral: Cognitive remediation
- Brain Training for Impaired Tone Matcher (Active Comparator): Cognitive remediation does not include sensory processing training
  Interventions: Behavioral: Cognitive remediation
- Brain Training for Intact Tone Matchers (Active Comparator): Cognitive remediation does not include sensory processing training
  Interventions: Behavioral: Cognitive remediation

INTERVENTIONS:
Behavioral: Cognitive remediation — Cognitive remediation sessions include working on computer based cognitive exercises and participating in a verbal discussion.

SUMMARY:
The purpose of this study is to develop and pilot test personalized and scalable approaches to Cognitive Remediation (CR) for schizophrenia and schizoaffective disorder. The intent is to more clearly define the therapeutic targets important to the facilitation of cognitive and functional improvement so that clinicians know how to customize cognitive interventions and deliver treatment in a more effective, efficient and personally relevant manner.

DETAILED DESCRIPTION:
There are three phases of this study.

Phase 1: Development and Adaptation. The goal of this phase is to adapt currently used computer based CR approaches to make them more personalized and scalable. We will create two CR interventions which differ in choice and pacing of the cognitive exercises. This phase is complete.

Phase 2: Open Trial and Intervention Refinement. The goal of this phase is to obtain quantitative and qualitative feedback on the acceptability and usability of the interventions from participants to inform further refinement of the assessment and treatment packages. We will recruit ten subjects from an outpatient psychiatric rehabilitation program in New York City. After determining study eligibility, individuals will complete a standardized neuropsychological battery for schizophrenia assessment, and a 5-minute Tone Matching Test to assess basic auditory processing. Participants will be randomly assigned to receive one of two intervention packages, developed in Phase 1. Each session includes 60 minutes of computer-based learning activities and a 15 minute therapist-led discussion that links the computer activities to cognition as applied to daily tasks and recovery goals. Participants will complete a total of 10 sessions attending 2-3 times weekly for 5 weeks. During each session, participants will be asked to keep a log of software used. At the conclusion of this abbreviated trial, the participants will participate in focus groups in which they will be asked to provide verbal feedback on how enjoyable, engaging, and useful they perceived the computer and discussion based exercises to be. Participants will be asked to provide verbal feedback on the assessment procedures. CR clinicians will join the research team to discuss participants' engagement and their experience with administering the Tone Matching Test and interventions. Qualitative data summarized from participant logs and focus groups will be considered by the research team to refine the assessment battery, treatment parameters, and rubric of learning exercises. This phase is complete.

Phase 3: Pilot Feasibility Trial. People with a diagnosis of schizophrenia or schizoaffective disorder may be referred by their treating clinician or may respond to posted advertisements to inquire about study participation. After being informed of study procedures, interested individuals will be asked to sign a consent form that documents willingness to participate in this study. Following informed consent, participants will be asked questions about demographic characteristics (e.g. age, education, employment), medication and psychosocial treatment status, psychiatric symptoms and symptoms severity, and will complete a brief assessment of estimated Intelligence. Those with an Intelligence Quotient (IQ) estimate below 70 or meeting substance dependence criteria at the time of evaluation will be exited from the study. In the same or second assessment session, participants will complete assessments of neuropsychological ability, current functioning, and motivation for treatment. Participants will then be randomly assigned to one of two treatment conditions named "Brain Basics" or "Brain Exercises".

Each treatment condition is structured in a group format of up to 5 participants. Both treatments use commercially available computer-based training software to exercise cognitive skills such as speed of processing, attention, working memory, and verbal memory. Both conditions will entail 50 minutes on the computer and 10 minutes group discussion. In the discussion, participants review the cognitive activities they are working on and how they will help them achieve their recovery goals. The treatment phase will consist of 30 separate sessions each 60 minutes in duration, administered 3 times a week over the course of a 10-week period. Participants will be re-tested on outcome measures approximately 1 week following end of treatment, and again 3 months later.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic and Statistical Manual-IV (DSM-IV) diagnosis of schizophrenia or schizoaffective disorder
2. Age 18 to 65
3. English speaking
4. Psychiatrically stable, verified by current living/treatment status

Exclusion Criteria:

1. Indication of mental retardation, determined by estimated IQ of less than 70
2. Hearing or visual impairment that precludes completing assessments
3. Neurologic illness that may affect brain physiology (e.g. Parkinson's, seizure disorder, epilepsy)
4. Current substance dependence symptoms in the past 6 weeks
5. Participation in cognitive remediation in the 12 months prior to study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2013-09; Primary Completion 2017-10-02 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Feasibility | Two years
  Feasibility of conducting a larger trial will be measured by recruitment, feasibility of enrollment, stratification, blinding and assessment, acceptability of randomization, retention of subjects

SECONDARY OUTCOMES:
Change in neurocognition from baseline to treatment end-point | 10 weeks
  Change in neurocognition will be measured with the MATRICS Consensus Cognitive Battery, including measures of: a) working memory; b) attention/vigilance; c) verbal learning; d) visual learning; e) processing speed; f) reasoning and problem solving.
Change in neurocognition from baseline to 3-month follow-up | 5.5 to 6 months
  Change in neurocognition will be measured with the MATRICS Consensus Cognitive Battery (see above).

OTHER OUTCOMES:
Tone Matching Ability - Treatment end-point | 10 weeks
  Tone matching (percent correct) will be assessed at baseline and at treatment end-point, using pairs of 100-ms tones in series, with 500-ms inter-tone interval.
UCSD Performance-Based Skills Assessment (UPSA)-Brief - treatment end-point | 10 weeks
  The UPSA - Brief is a proxy measure of daily functioning skills. Change from baseline to treatment end-point will be assessed.
Structured Clinical Interview for the Positive and Negative Syndrome Scale (SCI-PANSS) - Treatment end-point | 10 weeks
  The SCI-PANSS is a semi-structured interview containing 30 items that assess symptoms of psychotic disorders including positive, negative and general psychopathology. Change from baseline to treatment end-point will be assessed.
Intrinsic Motivation Inventory for Schizophrenia Research (IMI-SR) | 10 weeks
  Intrinsic Motivation Inventory for Schizophrenia Research (IMI-SR), a 21 item 7-point Likert type scale designed to assess a participant's subjective experience of an activity, specifically in an experimental setting (e.g. "I enjoyed doing this activity very much"). The IMI-SR will be administered at the first and last treatment sessions.
Perceived Competency Scale (PCS) | 10 weeks
  The PCS consists of 4 items on a 7-point Likert-type scale that assess feelings of competency when performing computer-based learning activities, with higher scores indicating greater perceived competency. The PCS will be administered at the first and last treatment sessions.
Tone Matching ability - 3-month follow up | 5.5 to 6 months
  Tone Matching (percent correct) will be assessed at baseline and 3-month follow-up, using pairs of 100-ms tones in series, with 500-ms inter-tone interval.
UCSD Performance-Based Skills Assessment (UPSA)-Brief - 3-month follow-up | 5.5 to 6 months
  The UPSA-Brief is a proxy measure for daily functioning skills. Change from baseline to 3-month follow-up will be assessed.
Structured Clinical Interview for the Positive and Negative Syndrome Scale (SCI-PANSS) - 3-month follow-up | 5.5 to 6 months
  The SCI-PANSS is a semi-structured interview containing 30 items that assess symptoms of psychotic disorders including positive, negative and general psychopathology. Change from baseline to 3-month follow-up will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Medalia, PhD, Principal Investigator — NYSPI
Locations (5):
- United States (5):
  - Williamsburg Clinic, Brooklyn, New York
  - Institute for Community Living, Brooklyn, New York
  - Nyspi/ Cumc, New York, New York
  - The Bridge Inc, New York, New York
  - FEGS Bronx Mental Health Clinic, The Bronx, New York

REFERENCES:
- [Result] Medalia A, Saperstein AM, Qian M, Javitt DC. Impact of baseline early auditory processing on response to cognitive remediation for schizophrenia. Schizophr Res. 2019 Jun;208:397-405. doi: 10.1016/j.schres.2019.01.012. Epub 2019 Jan 18. PMID 30665714